CLINICAL TRIAL: NCT04410627
Title: Pilot Trial Evaluating Usability, Acceptability, and Feasibility of the HoPE (Hospice Preparation and Education) Web-Based Tool
Brief Title: HoPE (Hospice Preparation and Education)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid/PI Vacancy
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00105058
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hospice Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Standard of Care + HoPE (Experimental)
  Interventions: Other: HoPE Website

INTERVENTIONS:
Other: HoPE Website — Educational website focused on hospice care
  Arms: Standard of Care + HoPE

SUMMARY:
The investigator will conduct a two-site, randomized, controlled study of the HoPE (Hospice Preparation and Education) web-based tool versus usual care to assess: Technology usability (primary), study feasibility (secondary), user acceptability (secondary), and hospice service conversion rate (exploratory). Technology usability will be assessed through a one-time quantitative survey using established instruments. Study feasibility and user accessibility will be assessed through trial enrollment and retention alongside analytics assessing tool usage (e.g. time spent on each page of the website). Conversion rate is the percent of patients introduced to hospice who eventually enroll. The investigators will evaluate in an exploratory manner the differential effect of HoPE versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for and referral made for home hospice services (Note: this excludes home palliative care, home infusion, home nursing, home physical therapy, and bridge services)
* Aged between 21 and 89
* Capacity to give consent
* Ability to speak and understand English

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Technology usability as measured by System Usability Scale | At study completion, up to 4 months.
  To determine usability, the System Usability Scale will be administered to each participant in the intervention arm. As described by usability.gov: "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking."

SECONDARY OUTCOMES:
Study Feasibility as measured by enrollment efficiency | At study completion, up to 4 months
  Enrollment efficiency will be measured by the percentage of patients approached who enroll in the study, with the goal of >50% enrollment.
Study Feasibility as measured by intervention completion | At study completion, up to 4 months
  Intervention completion will be measured by the percentage of participants on the intervention arm who complete at least 50% of the modules within the intervention website, with a goal of >50% of the participants.
User Accessibility as measured by Net Promoter score | At study completion, up to 4 months
  The Net Promoter scale is administered to participants in the intervention arm of the study only. This scale is an eleven-item likert scale assessing likelihood to recommend the intervention to a family member or friend. The percentage of participants who give a score of 0 through 6 is subtracted by the percentage of participants who give a score of 9 or 10 to give the overall Net Promoter score. This score is then compared to other scores of similar technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Kamal, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No